CLINICAL TRIAL: NCT04558216
Title: An Open-Label, Fixed-Sequence, Clinical Drug Interaction Study to Evaluate The Effect of a CYP3A-Inducer, Rifampin, on the Pharmacokinetics of Vonoprazan in Healthy Volunteers
Brief Title: Evaluation of Effect of Rifampin on the Pharmacokinetics of Vonoprazan in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to unavailability of rifampin for clinical trial use
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VONO-102
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Healthy Participants
Keywords: Vonoprazan; CYP3A; Rifampin
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vonoprazan single doses / rifampin single doses (Experimental): Participants will be administered a single oral dose of 20 mg of vonoprazan oral tablets on Day 1 and Day 17. Participants will also be administered single daily doses of 600 mg rifampin oral capsules on Days 3 through 18.
  Interventions: Drug: Vonoprazan; Drug: Rifampin

INTERVENTIONS:
Drug: Vonoprazan — 20 mg tablets administered orally
Drug: Rifampin — 600 mg (Two 300 mg capsules)

SUMMARY:
The primary objective of this study is to assess the effect of multiple doses of rifampin on the pharmacokinetics of vonoprazan in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Inclusion Criteria:

1. The participant is male or female 18 to 45 years of age, inclusive, at Screening.
2. The participant has a BMI 18 to 30 kg/m^2, inclusive, and has a body weight greater than 50 kg at Screening.
3. The participant is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at Screening.
4. Female participants of childbearing potential who may be sexually active with a non sterilized male partner must use an acceptable method of birth control (ie, diaphragm with spermicide, intrauterine device, condom with foam or vaginal spermicide, oral contraceptives, or abstinence) from the signing of informed consent until 4 weeks after the last dose of study drug or be surgically sterile (ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or postmenopausal (defined as amenorrhea for 12 consecutive months and documented plasma folical stimulating hormone [FSH] level >40 IU/mL).
5. Female participants must have a negative pregnancy test at Screening and Check-in.
6. The participant agrees to comply with all protocol requirements.
7. The participant is able to provide written informed consent.

Exclusion Criteria:

1. The participant has a history of any clinically significant neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urological, hematological, or endocrine disease or other abnormality that may affect the ability of the participant to participate in the study.
2. The participant has a positive test result for coronavirus disease 2019 (COVID-19), hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus type 1 or 2 antibodies at Screening.
3. The participant has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × the upper limit of normal (ULN) or total bilirubin >1.5 × ULN (with the exception of Gilbert's syndrome) at Screening or Check-in.
4. The participant has serum creatinine >1.2 mg/dL or blood urea nitrogen >20 mg/dL at Screening or Check-in.
5. The participant has any acute laboratory abnormality at Screening that precludes participation in the study, in the opinion of the investigator.
6. The participant has a current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome and asymptomatic gallstones).
7. The participant has used any prescription (excluding hormonal birth control) or over the counter medications (including CYP3A4 inducers) except paracetamol (up to 2 g per day), including herbal or nutritional supplements, within 14 days (or 5 half-lives) before the first dose of study drug or throughout the study.
8. The participant has consumed grapefruit or grapefruit juice, Seville orange or Seville orange containing products (eg, marmalade), or other food products that may be CYP3A4 inhibitors (eg, vegetables from the mustard green family [kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard] and charbroiled meats) within 7 days (or 5 half-lives) before the first dose of study drug or throughout the study.
9. The participant has consumed caffeine- or xanthine containing products within 48 hours (or 5 half lives) before the first dose of study drug or throughout the study.
10. The participant is a smoker or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 6 months before the first dose of study drug.
11. The participant has a history of alcohol abuse or drug addiction within the last year, excessive alcohol consumption (regular alcohol intake >21 units per week for male participants and >14 units of alcohol per week for female participants; 1 unit is equal to approximately 1/2 pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits), or use of alcohol 48 hours before the first dose of study drug or throughout the study.
12. The participant has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at Screening or Check-in.
13. The participant is involved in strenuous activity or contact sports within 24 hours before the first dose of study drug or throughout the study.
14. The participant has donated blood or blood products >450 mL within 30 days before the first dose of study drug.
15. The participant has a history of relevant drug and/or food allergies (ie, allergy to rifampin, vonoprazan, or excipients, or any significant food allergy that could preclude a standard diet in the clinical unit).
16. The participant has received study drug in another investigational study within 30 days of dosing.
17. Female participant is pregnant or lactating, intends to become pregnant before, during, or within 4 weeks after participating in this study, or intends to donate ova during this time period.
18. In the opinion of the investigator, the participant is not suitable for entry into the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-02-07 (Estimated); Study Completion 2021-02-19 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve from Time 0 to the Last Quantifiable Concentration (AUC0-t) of Vonoprazan | Day 1 and Day 17: 0.25 hours pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours post-dose
Area Under the Plasma Concentration Versus Time Curve from Time 0 Extrapolated to Infinity (AUC0-inf) of Vonoprazan | Day 1 and Day 17: 0.25 hours pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours post-dose
Maximum Observed Plasma Concentration (Cmax) of Vonoprazan | Day 1 and Day 17: 0.25 hours pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 30, 36, and 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Phathom Pharmaceuticals
Locations (1):
- PPD Development, LP, 7551 Metro Center Drive, Suite 200, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No